CLINICAL TRIAL: NCT01285895
Title: Assessing of the Educational Needs of Patients Who Received a Lung Transplantation or a Simultaneous Heart-lung Transplantation for Mucoviscidosis
Brief Title: Needs in Education for Pulmonary or Cardiopulmonary Transplanted Cystic Fibrosis Patients
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PROG/10/90
Record Dates: First submitted 2011-01-27; First posted 2011-01-28 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Cystic Fibrosis
Keywords: Lung and heart transplantations; Mucoviscidosis; Educational needs
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Main objective : This project aims to assess the educational needs of patients who received a lung transplantation or a simultaneous heart-lung transplantation for mucoviscidosis.

Specific objectives : Evaluate the specific needs dependent on seniority transplantation : 3 to 6 months, 6 months to 2 years, more than 2 years after transplantation

Secondary objectives :

* Assess the state of health
* Assess the knowledge
* Assess gestural know-how
* Assess the cognitive know-how
* Assess the behaviour adopted in reality by the patient
* Assess motivation psychosocial factors of :

  * self-efficacy and inefficiency
  * representation of obstacles, disadvantages of treatment
  * sense of control over their health
  * feeling of being supported by health professionals, by his close
  * representation of his responsibility to take care of his health, to follow his treatment, to be active about his treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients who received a lung transplantation or a simultaneous heart-lung transplantation for mucoviscidosis

Exclusion Criteria:

* Patient with a psychiatric disorder
* Patient in intensive care
* Palliative patient
* Patient aged under 18 years old
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received a lung transplantation or a simultaeous heart-lung transplantation for mucoviscidosis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valérie DAVID, Doctor, Principal Investigator — Nantes University Hospital; Romain GUILLEMAIN, Profesor, Study Chair — Hôpital Européen Georges-Pompidou; Jean-François MORNEX, Profesor, Study Chair — Hospices Civils de Lyon; Marc STERN, Profesor, Study Chair — Hôpital Foch; Martine REYNAUD-GAUBERT, Profesor, Study Chair — CHU de Marseille; Marlène MURRIS-ESPIN, Doctor, Study Chair — University Hospital, Toulouse; Romain KESSLER, Profesor, Study Chair — CHU de Strasbourg
Locations (1):
- Nantes University Hospital, Nantes, France